CLINICAL TRIAL: NCT06352762
Title: The Effects of Upper Extremity Robotic Rehabilitation on Upper Extremity Skills and Functional Independence Level in Patients With Spastic Hemiparetic Cerebral Palsy
Brief Title: The Effects of Upper Extremity Robotic Rehabilitation in Children With Spastic Hemiparetic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Nuriye BUYUKTAS, The Effects of Upper Extremity Robotic Rehabilitation in Children with Spastic Hemiparetic Cerebral Palsy, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Izmir Dokuz Eylul University
Record Dates: First submitted 2024-03-26; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Spastic Hemiplegic Cerebral Palsy; Upper Extremity Paresis; Robotic Rehabilitation
Keywords: Spastisity; Motor Function; Cerebral Palsy; Upper Extremity
MeSH Terms: conditions — Paresis; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study was conducted as a randomized controlled study.The first of the cases that met the study criteria was included in the study group, and the second in the control group. Randomization continued in this way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physiotherapy (Active Comparator): Strengthening and stretching exercises for lower and upper extremity muscles, hip and trunk stabilization training, balance training, gait training, upper extremity functional skills training, endurance training and coordination training were given.
  Interventions: Other: Conventional physiotherapy
- Robotic Rehabilitation (Experimental): Strengthening and stretching exercises for lower and upper extremity muscles, hip and trunk stabilization training, balance training, gait training, upper extremity functional skills training, endurance training and coordination training were given. In addition, upper extremity robotic rehabilitation was applied.
  Interventions: Other: Robotic Rehabilitation

INTERVENTIONS:
Other: Conventional physiotherapy — Strengthening and stretching exercises for lower and upper extremity muscles, hip and trunk stabilization training, balance training, gait training, upper extremity functional skills training, endurance training and coordination training were given. Exercises were planned according to the developmental stage. Sessions were applied 3 days a week and 45 minutes for 5 weeks, for a total of 15 sessions.
  Arms: Conventional physiotherapy
Other: Robotic Rehabilitation — Strengthening and stretching exercises for lower and upper extremity muscles, hip and trunk stabilization training, balance training, gait training, upper extremity functional skills training, endurance training and coordination training were given. Exercises were planned according to the developmental stage. Sessions were applied 3 days a week and 45 minutes for 5 weeks, for a total of 15 sessions. An additional 30 minutes of robotic rehabilitation was applied to the conventional physiotherapy program. Robotic rehabilitation was applied after each session of conventional physiotherapy applications.
  Arms: Robotic Rehabilitation

SUMMARY:
Aims: To investigate the effects of upper extremity robotic rehabilitation on upper extremity skills and functional independence level in patients with hemiparetic Cerebral Palsy (hCP).

Methods: 34 hCP patients attended the study. 17 children in the training group recived conventional physiotherapy and Robotic Rehabilitation. 17 children in the control group recived only conventional physiotherapy. Convantional physiotherapy program lasted 45 minutes, Robotic Rehabilitation program lasted 30 minutes. All participants were enrolled in sessions 3 times a week for 5 weeks. Measurements were made before and after the therapy. Outcome measures were Modified Ashworth Scale (MAS) for muscle tone, Abilhand-Kids Test for manual skills, The Quality of Upper Extremity Skills Test (QUEST) for upper extremity motor function and The WeeFIM for functional independence level.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a permanent but non-progressive neurodevelopmental disorder that occurs in the immature brain and causes activity limitations in children. Epilepsy, cognitive disorders, behavioral disorders, visual-hearing losses and sensory disorders may be observed in children with CP along with motor damage. Motor dysfunction disorders constitute one of the most basic problems in patients with CP. Hand-arm coordination disorders, grip disorders and sensory disorders in the upper extremities negatively affect the daily life activities and functional independence levels of patients. It has been shown that neglect occurs with advancing age in cases with CP when upper limb treatment is delayed, and compensation mechanisms develop involving the use of unaffected side upper limbs to ensure daily living activities. Upper limb functional skills are very important to be able to perform daily life activities. It is not possible to perform activities such as holding and releasing objects, reaching for objects with non-functional upper limbs. Abnormal posture and deformities caused by spasticity restrict the functions of the upper extremities, make daily living activities difficult and increase the burden of people caring for the child. With the technological developments in recent years, virtual reality applications and robotic rehabilitation programs play an important role in CP rehabilitation. Significant improvements have been shown, especially in the development of walking, balance and postural control. Intensive practical, frequent repetitive movements and functional activities can be provided simultaneously in the same session with robotic rehabilitation applications. In the literature, the effects of robotic rehabilitation applications have been investigated in adult neurological patients. In pediatric patients, studies generally focus on lower limb function and walking. The number of studies examining the effect of robotic rehabilitation on upper limb functions in children with CP are limited. Based on these deficiencies in the literature, the purpose of the planned study was to examine the effect of upper limb robotic rehabilitation on upper limb functions and functional independence level in children diagnosed with spastic hemiparetic CP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spastic hemiparetic CP
* Upper extremity muscle tone between 1-3 according to the Modified Ashworth Scale
* According to Gross Motor Functional Clasification System level 1-2-3
* Able to understand simple instructions

Exclusion Criteria:

* Having a history of epilepsy
* Having botox in the last 6 months
* Having surgery in the last 6 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Muscle Tone | Assessment was performed twice, before treatment started and at the end of the fifth week.
  Muscle tone was assessed using the Modified Ashworth Scale. Resistance to passive movement was scored from 0 to 5. Higher scores indicate higher muscle tone. Shoulder extensors, adductors and internal rotators; elbow flexors; forearm pronators, wrist and finger flexors were evaluated. Each region was evaluated individually, and the sum of the measured regions was calculated to determine overall muscle tone.
Upper Extremity Motor Function | Assessment was performed twice, before treatment started and at the end of the fifth week.
  The Quality of Upper Extremity Skills Test (QUEST) was used. The test evaluates dexterity and quality of movement. It consists of a total of 7 headings (Independent movements, grasping, weight bearing, protective extension, degree of hand function, degree of spasticity, level of cooperation) and 34 items. Each item is scored between 0-2. A score of 0 indicates that the movement was not achieved, 1 point indicates that it was partially achieved, and 2 points indicates that it was completely achieved. High scores from the test indicate good upper extremity motor functions.
Manual Ability | Assessment was performed twice, before treatment started and at the end of the fifth week.
  Abilhand-Kids test was used. This test evaluates children's abilities in daily living activities for the hand and upper extremity. The test consists of 21 items. Each item is scored between 0-2. A score of 0 means that the activity cannot be done, a score of 1 means that the child has difficulty in doing the activity, and a score of 2 means that the activity can be done easily. High scores from the test indicate good manual abilities.
Functional Independence | Assessment was performed twice, before treatment started and at the end of the fifth week.
  It was assessed using the pediatric functional independence scale (WeeFIM). It contains a total of 6 topics and 18 questions, including self-control, sphincter control, transfers, locomotion, communication, social and cognitive functions. Each item is scored between 1-7. High scores from the test indicate a high level of independence.

CONTACTS AND LOCATIONS:
Overall Officials: Nuriye Büyüktaş, MsC, Principal Investigator — Izmir Bakircay University
Locations (1):
- Nuriye Büyüktaş, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No